CLINICAL TRIAL: NCT05621265
Title: Efficacy of Automated Text Messaging Services on Sleep Health, Stress, Pain, and Function in Physical Therapy Patients
Brief Title: Efficacy of Automated Text Messaging Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Black Hills State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BlackHillsSTATE
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Physical Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Automated Text messaging for sleep behavior change
  Interventions: Behavioral: Automated Text messaging
- Control (No Intervention): Control, Traditional physical therapy only

INTERVENTIONS:
Behavioral: Automated Text messaging — daily text message
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test automated text messaging as an effective behavior change intervention in physical therapy patients. The main purpose of this study was to trial sleep hygiene education for improving physical therapy patients' sleep through the use of daily automated text messaging. Researchers will compare two groups to see if the intervention group which consisted of participants getting daily automated text messages for sleep hygiene tips would be effective in improving sleep, health, pain, and function compared to a group that is receiving traditional physical therapy alone.

DETAILED DESCRIPTION:
Participants will be recruited from the outpatient physical therapy clinic verbally by their therapist and by an informational handout they receive from the therapist. The student researcher (who also works at this clinic) will then contact the participant to set up a time to complete the initial survey questions at the clinic in a private treatment room. During the initial visit, participants will read through and sign informed consent explaining the procedures and expectations of them during the study. The participants will then complete the following questionnaires: Pittsburgh Sleep Quality Index, Sleep Hygiene Index, Medical Outcome Survey-sleep 9, Perceived Stress Scale, Numeric Pain Rating Scale, and Patient Specific Functional Scale. The participants will randomly be assigned to one of two groups. The intervention group will receive daily automated text messages scheduled for 8:00 pm every evening. The text messages will include a variety of sleep hygiene behavioral tips for the participant to try. This will last for a total of four weeks. The control group will not receive any intervention during this time frame. Following the four weeks, student researchers will return to each participant's clinic to collect the same data that was collected at the initial visit. Each participant will have a total of 2 sessions to complete with each session taking approximately 15-30 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

Adults 18 years and older seeking outpatient Physical Therapy

Exclusion Criteria:

Inability to access a smart-phone or computer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | initial visit and 4-week follow up
  sleep quality measurement. Scores range 0-21 with higher score indicating poorer sleep quality.
Sleep Hygiene Index | initial and 4-week follow up
  measuring participants sleep hygiene behaviors. Scores range 0-52 with a higher score indicating poorer sleep hygiene.

SECONDARY OUTCOMES:
Perceived Stress Scale | initial and 4-week follow up
  stress measurement. Scores range 0-40 with higher score indicating greater stress.
Patient Specific Functional Scale | initial and 4-week follow up
  scale for improving patient's top three chosen functions they want to improve. Scores range from 0-10 with lower scores indicating poorer function.
Numeric Pain rating Scale | Initial and 4-week follow up
  tool to measure pain. 0-10 with 10 being highest pain possible.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Pfeiffer, DPT, Principal Investigator — Black Hills State University
Locations (1):
- Black Hills Physical Therapy, Spearfish, South Dakota, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share all data from excel.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data is available now for anyone who is interested.
Access Criteria: Data will be available by request through emailing the PI Ashley Pfeiffer at ashley.pfeiffer@bhsu.edu